CLINICAL TRIAL: NCT00625274
Title: A Randomized, Open-Label, Comparative 3-Way Treatment Crossover Study of 24-Hour Intragastric pH Profile of Once Daily Oral Administration of Esomeprazole 40mg, Lansoprazole 30mg, and Pantoprazole 40mg at Steady State in NSAID-Using Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Tore Lind, MD - Nexium Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D9612L00063
Record Dates: First submitted 2008-02-20; First posted 2008-02-28 (Estimated); Last update posted 2008-02-28 (Estimated); Status verified 2008-02

CONDITIONS: Heartburn; Upper Abdominal Pain; Nausea; Acid Regurgitation
Keywords: Nexium; esomeprazole; lansoprazole; pantoprazole; Nonsteroidal Anti-Inflammatory Drugs (NSAIDs)
MeSH Terms: conditions — Heartburn; Abdominal Pain; Nausea | interventions — Esomeprazole; Lansoprazole; Pantoprazole

ARMS (3):
- 1 (Experimental): Oral
  Interventions: Drug: Esomeprazole
- 2 (Experimental): Oral
  Interventions: Drug: Lansoprazole
- 3 (Experimental): Oral
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Esomeprazole — 40mg Oral
  Other Names: Nexium
  Arms: 1
Drug: Lansoprazole — 30mg Oral
  Other Names: Prevacid
  Arms: 2
Drug: Pantoprazole — 40mg Oral
  Other Names: Protonix
  Arms: 3

SUMMARY:
This study looks at controlling intragastric pH following administration of esomeprazole 40 mg, lansoprazole 30 mg and pantoprazole 40 mg taken orally, once daily in patients taking either non-selective or cyclooxygenase-2 (COX-2) selective nonsteroidal anti-inflammatory drugs (NSAIDs).

ELIGIBILITY:
Inclusion Criteria:

* A medical diagnosis of a condition that requires daily Nonsteroidal Anti-Inflammatory Drugs (NSAID) treatment for at least 5 days per week for 1 month prior to entering the study and during the study.
* Some patients will need to undergo an upper endoscopy at screening.

Exclusion Criteria:

* Signs of clinically significant (GI) bleeding (e.g., melena, frank hematochezia) at the time of the baseline EGD or within 3 days prior to randomization.
* History of gastric or esophageal surgery (including but not limited to Nissen fundoplication, bariatric surgery (e.g. gastric stapling or Roux-En-Y gastric bypass), vagotomy, or Billroth operation).
* Many further exclusion criteria, please refer to the investigator site.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2004-06; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
To compare the pharmacodynamic efficacy in controlling intragastric pH (percent time pH > 4.0) following administration of esomeprazole 40 mg, lansoprazole 30 mg and pantoprazole 40 mg taken orally, once daily in pat | Screening, assessments every 2 weeks.

SECONDARY OUTCOMES:
To compare nocturnal intragastric acid control in NSAID-using patients taking esomeprazole 40 mg, lansoprazole 30 mg or pantoprazole 40 mg once daily. | Patients will be an in-patient beginning the AM of Day 5 through the AM of Day 6 during all three treatment periods.
To compare intragastric acid control utilizing thresholds other than pH 4.0 among NSAID-using patients taking esomeprazole 40 mg, lansoprazole 30 mg and pantoprazole 40 mg once daily. | Patients will be an in-patient beginning the AM of Day 5 through the AM of Day 6 during all three treatment periods.
To compare the mean hourly cumulative integrated gastric acidity during the 24-hour monitoring period on Day 5 among NSAID-using patients taking esomeprazole 40 mg, lansoprazole 30mg and pantoprazole 40 mg once daily. | 24-hour monitoring period

CONTACTS AND LOCATIONS:
Overall Officials: Paula Fernstrom, Study Director — Nexium Global Product Director, AstraZeneca